CLINICAL TRIAL: NCT06651281
Title: A Phase 3 Extension Study to Evaluate the Long-term Safety and Efficacy of Tulisokibart in Participants With Crohn's Disease or Ulcerative Colitis
Brief Title: Extension Study of Long-term Safety and Efficacy of Tulisokibart in Participants With Crohn's Disease or Ulcerative Colitis (MK-7240-011)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7240-011; 2024-513533-20-00 (Registry Identifier: EU CT); U1111-1306-6970 (Registry Identifier: UTN)
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Crohn Disease; Colitis, Ulcerative
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: This extension study will enroll participants who choose to enter from certain studies in which they are already receiving treatment (their "parent studies"). They will enter the appropriate arm in this study that will provide the same treatment they had been receiving on their parent study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants in "Group 1: Low Dose Unblinded" and "Group 2: High Dose Unblinded" received open-label treatment on their parent studies, and will remain unblinded on this extension study.
  Participants in "Group 3: High Dose Blinded" and "Group 4: Low Dose Blinded" were all blinded on their parent studies, and will remain blinded on this extension study until after regulatory approval or market authorization in the United States or European Medicines Agency, per sponsor discretion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: Low Dose Unblinded (Experimental): Participants receive a low dose subcutaneous (SC) tulisokibart regimen.
  Interventions: Drug: Tulisokibart
- Group 2: High Dose Unblinded (Experimental): Participants receive a high dose SC tulisokibart regimen.
  Interventions: Drug: Tulisokibart
- Group 3: High Dose Blinded (Experimental): Participants receive a blinded high dose SC tulisokibart regimen.
  Interventions: Drug: Tulisokibart
- Group 4: Low Dose Blinded (Experimental): Participants receive a blinded low dose SC tulisokibart regimen.
  Interventions: Drug: Tulisokibart; Drug: Placebo to tulisokibart

INTERVENTIONS:
Drug: Tulisokibart — Humanized monoclonal antibody that binds human tumor necrosis factor-like cytokine 1A (TL1A), administered subcutaneously
  Other Names: MK-7240
Drug: Placebo to tulisokibart — Placebo matching SC tulisokibart
  Arms: Group 4: Low Dose Blinded

SUMMARY:
Researchers want to learn more about tulisokibart (also known as MK-7240) in an extension study. Tulisokibart is a medicine designed to treat active, moderate to severe Crohn's disease (CD) and ulcerative colitis (UC). An extension study is a type of study where people who received tulisokibart in certain other studies for CD or UC (called a parent study) may be able to join this study. The goals of this study are to learn about the safety of tulisokibart over time in people with CD or UC, and if people tolerate it.

ELIGIBILITY:
Inclusion Criteria:

* Has participated in a qualifying tulisokibart Phase 2 or Phase 3 parent study for CD or UC
* The investigator determines that the participant derives clinical benefit from continued study intervention based upon clinical evaluations performed during their parent study
* A participant assigned female sex at birth is not breastfeeding during the study intervention period and for at least 14 weeks after the last dose of study intervention
* A participant of childbearing potential (POCBP) is not pregnant and has a negative highly sensitive pregnancy test (urine or serum) as required by local regulations within 24 hours (for a urine test) or 72 hours (for a serum test) before the first dose of study intervention
* A POCBP uses an acceptable contraceptive method, or adheres to penile-vaginal intercourse abstinence as their preferred and usual lifestyle (abstinent on a long-term and persistent basis)

Exclusion Criteria:

* Has prematurely discontinued study intervention in their parent study
* Has received any protocol-specified prohibited medications during their parent study
* Has known allergies, hypersensitivity, or intolerance to tulisokibart or its excipients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1380 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2037-12-17 (Estimated); Study Completion 2037-12-17 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 378 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 364 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment due to an AE will be reported.

SECONDARY OUTCOMES:
Percentage of Participants with Crohn's Disease Achieving Clinical Remission per Crohn's Disease Activity Index (CDAI) Score | Week 364
  The percentage of participants who enrolled in their parent study with Crohn's disease who achieve clinical remission, as defined by CDAI score <150, at Week 364 will be presented.
Percentage of Participants with Crohn's Disease Achieving Clinical Remission per Stool Frequency and Abdominal Pain Score | Week 364
  The percentage of participants who enrolled in their parent study with Crohn's disease achieving clinical remission at Week 364 per stool frequency/abdominal pain score (SF/APS), as defined by average daily SF ≤2.8 and average daily APS ≤1.0 and both not greater than baseline will be presented.
Percentage of Participants with Crohn's Disease With Endoscopic Remission Per Simplified Endoscopic Score for Crohn's Disease (SES-CD) | Week 364
  The Simplified Endoscopic Score for Crohn's Disease (SES-CD) measures ileocolonoscopic findings in Crohn's Disease. Each segment of the ileo-colon (terminal ileum; ascending, transverse, and descending colon; rectum) is scored from 0 (normal or inactive disease) to 12 (severe disease; no more than one segment can have a score of 12, in which case the other 4 segments must each be ≤11), and the scores summed to produce an SES-CD ranging from 0 (overall least severe disease) to 56 (overall most severe disease). Endoscopic remission is defined as an SES-CD ≤4 and at least 2-point reduction from baseline and no subscore >1 in any individual variable, as scored by central reader.
Percentage of Participants with Ulcerative Colitis Achieving Clinical Remission Per Modified Mayo Score (MMS) | Week 364
  The Modified Mayo Score (MMS) is a composite score of ulcerative colitis (UC) disease activity on a scale of increasing severity from 0-9, calculated by summing three subscores: Endoscopic subscore (ES), scored on a scale of increasing severity from 0 (normal or inactive disease) to 3 (severe disease, such as spontaneous bleeding or ulceration); Stool frequency subscore (SFS), scored on a scale of increasing frequency from 0 (normal number of stools) to 3 (≥5 stools more than normal per day for the participant); and rectal bleeding subscore (RBS), scored on a scale of increasing severity from 0 (no blood seen) to 3 (blood alone passed). Clinical Remission is defined as an ES of 0 or 1, RBS of 0, and SFS of 0 or 1 and not greater than the baseline SFS.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (37):
- United States (12):
  - Connecticut Clinical Research Institute ( Site 0297), Bristol, Connecticut
  - St. Joseph Mercy Hospital - Huron Gastroenterology Associates ( Site 0287), Ypsilanti, Michigan
  - BVL Research - Kansas ( Site 0292), Liberty, Missouri
  - New York Gastroenterology Associates ( Site 0253), New York, New York
  - GI Alliance - Digestive Health Associates of Texas - DHAT ( Site 0290), Garland, Texas
  - GI Alliance - Lubbock ( Site 0288), Lubbock, Texas
  - Caprock Gastro Research ( Site 0293), Lubbock, Texas
  - Southern Star Research Institute ( Site 0299), San Antonio, Texas
  - GI Alliance - Southlake ( Site 0298), Southlake, Texas
  - Tyler Research Institute ( Site 0294), Tyler, Texas
  - University of Virginia Health System ( Site 0291), Charlottesville, Virginia
  - Washington Gastroenterology - Tacoma ( Site 0295), Tacoma, Washington
- Czechia (2):
  - Vojenská Nemocnice Brno-Internal department ( Site 0701), Brno, Brno-mesto
  - Hepato-Gastroenterologie HK ( Site 0700), Hradec Králové
- France (4):
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet ( Site 1002), Nice, Alpes-Maritimes
  - CMC Ambroise Paré Hartmann - Institut des MICI ( Site 1003), Neuilly-sur-Seine, Hauts-de-Seine
  - CHRU De Nancy - Hopital de Brabois ( Site 1001), Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Hopital Claude Huriez CHRU LILLE ( Site 1004), Lille, Nord
- ARENSIA Exploratory Medicine Georgia ( Site 1104), Tbilisi, Georgia
- Hungary (2):
  - Békés Megyei Központi Kórház Dr. Réthy Pál Tagkórház-4. Belgyogyaszat Gasztroenterologia ( Site 1411), Békéscsaba, Bekes County
  - Semmelweis Egyetem ( Site 1400), Budapest
- Poland (14):
  - Rivermed Sp. z.o.o. ( Site 2206), Poznan, Greater Poland Voivodeship
  - Centrum Diagnostyczno - Lecznicze Barska sp. z o.o. ( Site 2208), Włocławek, Kuyavian-Pomeranian Voivodeship
  - Krakowskie Centrum Medyczne ( Site 2210), Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne Oporow ( Site 2212), Wroclaw, Lower Silesian Voivodeship
  - Melita Medical ( Site 2204), Wroclaw, Lower Silesian Voivodeship
  - Przychodnia Futuremeds Wroclaw ( Site 2211), Wroclaw, Lower Silesian Voivodeship
  - 1 Wojskowy Szpital Kliniczny Z Poliklinika SPZOZ w Lublinie ( Site 2205), Lublin, Lublin Voivodeship
  - Medrise Sp. z o.o. ( Site 2200), Lublin, Lublin Voivodeship
  - Centrum Zdrowia MDM ( Site 2202), Warsaw, Masovian Voivodeship
  - Vivamed Sp. z o.o. ( Site 2201), Warsaw, Masovian Voivodeship
  - WIP Warsaw IBD Point Professor Kierkus ( Site 2209), Warsaw, Masovian Voivodeship
  - Vita Longa Sp. Zoo ( Site 2213), Katowice, Silesian Voivodeship
  - Sonomed Sp. z o. o. ( Site 2203), Szczecin, West Pomeranian Voivodeship
  - Bonifraterskie Centrum Medyczne ( Site 2207), Lodz, Łódź Voivodeship
- United Kingdom (2):
  - Whipps Cross University Hospital ( Site 3400), London, England
  - MAC Research - Merseyside ( Site 3401), Prescot, Knowsley

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26142&tenant=MT_MSD_9011